CLINICAL TRIAL: NCT05170958
Title: A Phase I/II Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetic Characteristics and Preliminary Efficacy of LBL-024 in Patients With Advanced Malignant Tumors
Brief Title: A Phase I/II Clinical Study of LBL-024 in Patients With Advanced Malignant Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nanjing Leads Biolabs Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LBL-024-CN001
Record Dates: First submitted 2021-11-17; First posted 2021-12-28 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LBL-024 (Experimental): LBL-024 injection; Initial dose - MTD; Q3W
  Interventions: Drug: LBL-024 for Injection

INTERVENTIONS:
Drug: LBL-024 for Injection — LBL-024 was given every three weeks for treatment
  Other Names: LBL-024

SUMMARY:
To evaluate the phase I/II clinical study of LBL-024 in the treatment of patients with advanced malignant tumors

DETAILED DESCRIPTION:
This trial is a single-arm, open-label, phase I/II clinical study of LBL-024 in patients with advanced malignant tumors. The phase I dose escalation and PK expansion phase plans to include patients with advanced malignant tumors who have failed previous standard treatment or do not have standard treatment or are not applicable to standard treatment at this stage. The phase IIa indication expansion phase plans to include patients with advanced malignant tumors , and evaluate the safety, tolerability, pharmacokinetic (PK) characteristics, immunogenicity and preliminary efficacy. Single-arm registry clinical study to be conducted in Phase IIb.

This trial includes two parts:

Part I: A Phase I/IIa clinical study on the safety, tolerability, PK and efficacy of LBL-024 in patients with advanced malignant tumor.

Part II:Phase IIb is a pivotal single-arm clinical study.

ELIGIBILITY:
Inclusion Criteria:

1. Agree to comply with the trial treatment plan and visit plan, voluntarily agree to sign the informed consent form;
2. 18-75 years old (including boundary value), no gender limit in the I/IIa trial phase；18-80 years old (including boundary value), no gender limit in the IIb trial phase；
3. Subject has adequate organ and bone marrow function，Conforming to laboratory test results:
4. The expected survival time is at least 12 weeks
5. ECOG score is 0-1
6. Males with fertility and females of childbearing age are willing to take effective contraceptive measures From the signing of the informed consent form to within 6 months after the last administration of the trial drug (including abstinence, intrauterine device, various hormonal contraception, correct use of contraception Sets，etc）; Women of childbearing age include pre-menopausal women and women within 2 years after menopause. Women of childbearing age must have a negative pregnancy test within 7 days before the first trial drug is administered.

Exclusion Criteria:

1. Receiving other unmarketed clinical research drugs or treatments within 4 weeks before using the research drug for the first time;
2. Brain parenchymal metastases or meningeal metastases with clinical symptoms, which are not suitable for inclusion in the group by the investigator's judgment;
3. medical history of immunodeficiency including positive HIV antibody test;
4. Women who are pregnant or breastfeeding;
5. The investigator believes that the subject has other conditions that may affect compliance or are not suitable for participating in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 396 (Estimated)
Dates: Start 2022-01-06 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | All subjects signed the informed consent form to the completion of the follow-up period of drug withdrawal （Visit 30 days after discontinuation of treatment or withdraw from the visit）
  During the dose-escalation phase, the highest dose of dose-limiting toxicity for subjects less than or equal to 1/6 of the study drug within 3 weeks of starting treatment in Phase I study.
Dose-limiting toxicities（DLT) | Within 3 weeks after receiving the first dose of the test drug
  During the DLT observation period, the subject has an event that is reasonably related to the test drug (possibly, likely or definitely related) in Phase I study.
Objective Response Rate (ORR) | All subjects signed the informed consent form to the completion of the follow-up period of drug withdrawal （Visit 30 days after discontinuation of treatment or withdraw from the visit）
  Defined as the percentage of subjects having a Complete Response or Partial Response(ORR, including after immunotherapy complete response (iCR) and partial response (iPR)),will be determined by investigator assessment of radiographic disease assessments per RECIST V1.1. It was used to evaluate the efficacy of LBL-024 in Phase II study.

SECONDARY OUTCOMES:
Adverse events and serious adverse events | All subjects signed the informed consent form to the completion of the follow-up period of drug withdrawal （Visit 30 days after discontinuation of treatment or withdraw from the visit）
  Laboratory examination, physical examination, vital signs and electrocardiogram, etc.
Maximum serum concentration (Cmax) | All subjects signed the informed consent form to the completion of the follow-up period of drug withdrawal （Visit 30 days after discontinuation of treatment or withdraw from the visit）
  To determine the PK profile of LBL-024
Immunogenicity | All subjects signed the informed consent form to the completion of the follow-up period of drug withdrawal （Visit 30 days after discontinuation of treatment or withdraw from the visit）
  Incidence of subjects with anti-drug antibody (ADA) and neutralizing antibody (if applicable)
Disease Control Rate(DCR) | Visit 30 days after discontinuation of treatment or withdraw from the visit
  Defined as percentage of participants having CR, PR, iCR，iPR or SD as best on-study response
Progression-free survival (PFS) | All subjects signed the informed consent form to the completion of the follow-up period of drug withdrawal（Visit 30 days after discontinuation of treatment or withdraw from the visit）
  Defined as the time from random assignment in a clinical trial to disease progression or death from any cause, has recently become an endpoint of considerable interest in the study of new oncology drugs.

CONTACTS AND LOCATIONS:
Overall Officials: lin Shen, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (49):
- China (49):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Anhui Provincial Hospital, Hefei, Anhui
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Chongqing Cancer Hospital, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - The First Affiliated Hospital,Sun Yat-sen University, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guanzhou, Guangdong
  - Guangxi Medical University Cancer Hospital & Guangxi Cancer Institute, Nanning, Guangxi
  - Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou
  - Sir Run Run Shaw Hospital, Hangzhou, Hangzhou
  - Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Anyang Tumor Hospital, Anyang, Henan
  - The First Affilated Hospital of Henan University of Science & Technology, Luoyang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Tongji Hospital, Wuhan, Hubei
  - Wuhan Union Hospital of China, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Xiangyang Central Hospital, Xiangyang, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Nanjing First Hospital, Nanjing, Jiangsu
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - The Second Affiliated Hospital Nanchang University, Nanchang, Jiangxi
  - The Ferst Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Ch’ang-ch’un, Jilin
  - Liaoning Cancer Hospital & Institute, Shenyang, Liaoning
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Shandong Cancer Hospital & Institute, Jinan, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - Shanxi Provincial Cancer Hospital, Taiyuan, Shanxi
  - The First Affiliated Hospital of Xi'An Jiaotong University, Xi’an, Shanxi
  - Sichuan Cancer Hospital, Chengdu, Sichuan
  - Mianyang Central Hospital, Mianyang, Sichuan
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The First Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No